CLINICAL TRIAL: NCT02212197
Title: A Phase II, Open Label, Active Control, Multi-National, Multi-Centre, Randomized, Parallel Group Study Assessing Pharmacokinetics, Pharmacodynamics, Efficacy and Safety of CAM2032 (Leuprolide Acetate FluidCrystal® Injection Depot Once Monthly) After Repeat Doses of 3.75 mg and 7.5 mg of Leuprolide Acetate vs. Eligard® 7.5 mg in Patients With Prostate Cancer
Brief Title: Phase II Study of Subcutaneous Injection Depot of Leuprolide Acetate in Patient With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-12-460
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; leuprolide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAM2032 3.75 mg (Experimental): Single subcutaneous buttock injections of CAM2032 (leuprolide acetate FluidCrystal® injection depot) 3.75 mg on Days 0, 28 and 56.
  Interventions: Drug: leuprolide acetate FluidCrystal® injection depot
- CAM2032 7.5 mg (Experimental): Single subcutaneous buttock injections of CAM2032 (leuprolide acetate FluidCrystal® injection depot) 7.5 mg on Days 0, 28 and 56.
  Interventions: Drug: leuprolide acetate FluidCrystal® injection depot
- Eligard 7.5 mg (Active Comparator): Single subcutaneous buttock injections of Eligard® (leuprolide acetate) 7.5 mg on Days 0, 28 and 56.
  Interventions: Drug: leuprolide acetate

INTERVENTIONS:
Drug: leuprolide acetate FluidCrystal® injection depot
  Other Names: CAM2032
  Arms: CAM2032 3.75 mg; CAM2032 7.5 mg
Drug: leuprolide acetate
  Other Names: Eligard
  Arms: Eligard 7.5 mg

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, pharmacodynamics, efficacy and safety of CAM2032 versus Eligard, in patients with prostate cancer. All patients will receive leuprolide acetate administered subcutaneously once monthly during 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥40 and ≤85 years of age
* Histological or cytological proven adenocarcinoma of the prostate requiring hormone therapy
* Life expectancy over 12 months
* World Health Organisation/ The Eastern Cooperative Oncology Group (WHO/ECOG) performance status of 0, 1 or 2
* Adequate and stable renal function
* Adequate and stable hepatic function

Exclusion Criteria:

* Evidence of brain metastasis, spinal cord compression, or urinary tract obstruction
* Serum Testosterone levels below 150 ng/dL at Screening visit
* Medical or radiological prostate cancer treatments within 2 months prior to the Screening visit
* Surgical treatment of prostate cancer within 2 weeks prior to the Screening visit
* Prior orchiectomy, hypophysectomy, or adrenalectomy
* Prior use of LHRH agonists within 12 months prior to the Screening visit and during the study

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo Tammela, Prof, Principal Investigator — Tampere University Hospital
Locations (7):
- Finland (4):
  - Docrates Cancer Center, Helsinki
  - University Hospital of Helsinki, Department of Urology, Helsinki
  - Tampere University Hospital, Department of Urology, Tampere
  - University Hospital of Turku, Department of Urology, Turku
- Hungary (3):
  - Semmelweis University Hospital Department of Urology, Budapest
  - Szent Imre Teaching Hospital, Budapest
  - University of Debrecen, Medical Health Sciences Center, Department of Urology, Debrecen

RESULTS

PARTICIPANT FLOW:
Groups:
- Eligard 7.5 mg: Single subcutaneous buttock injections of Eligard® 7.5 mg on Days 0, 28 and 56.
Period: Overall Study
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Started | 19 | 15 | 17
Completed | 18 | 15 | 17
Not Completed | 1 | 0 | 0
Not completed — Need for radiotherapy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg | Total
Number analyzed (Participants) | 19 | 15 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 2 | 9
  >=65 years | 13 | 14 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.5) | 71.9 (6.3) | 70.9 (7) | 70.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 15 | 17 | 51
Region of Enrollment [Number; unit: participants]
  Hungary | 6 | 5 | 9 | 20
  Finland | 13 | 10 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Observed Maximum Serum Leuprolide Concentration (Cmax) for Dose 1 and Dose 3
Description: Blood samples for analysis of serum leuprolide concentrations were collected at pre-determined time points throughout the trial (with full PK profiles after Dose 1 and Dose 3). The PK parameter, Cmax was derived for Doses 1 and 3 of the investigational medicinal product (IMP).
Time Frame: 84 days
Population: The Per-Protocol Set (PPS) consisted of all randomized participants in the safety population who had a complete PK profile. In the CAM2032 3.75 mg group 15 of the 19 randomized participants were included in the PPS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
ng/mL
  Dose 1 | 6.14 (41.1) | 9.66 (31.5) | 13.6 (54.7)
  Dose 3 | 5.36 (33.3) | 11.3 (36.8) | 12.1 (47.3)

2. Primary Outcome: Apparent Terminal Half-life (t½) for Dose 1 and Dose 3
Description: Blood samples for analysis of serum leuprolide concentrations were collected at pre-determined time points throughout the trial (with full PK profiles after Dose 1 and Dose 3). The PK parameter, t1/2 was derived for Doses 1 and 3 of the IMP.
Time Frame: Days 0-28 and Days 56-84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
hour
  Dose 1 | 205 (113) | 231 (142) | 743 (1677)
  Dose 3 | 299 (277) | 434 (867) | 378 (570)

3. Primary Outcome: Area Under the Serum Concentration-time Curve (AUC) Over the Dosing Interval (AUCtau) for Dose 1 and Dose 3
Description: Blood samples for analysis of serum leuprolide concentrations were collected at pre-determined time points throughout the trial (with full PK profiles after Dose 1 and Dose 3). The PK parameter, AUCtau was derived for Doses 1 and 3 of the IMP.
Time Frame: Days 0-28 and Days 56-84 (0-672 hours after Doses 1 and 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
h*ng/mL
  Dose 1 | 329 (37.6) | 622 (45.2) | 397 (45.3)
  Dose 3 | 343 (24.7) | 757 (53.4) | 460 (62.2)

4. Secondary Outcome: Time (Days) to Testosterone Recovery After Dose 3
Description: The pharmacodynamic (PD) effects of leuprolide were assessed by measuring serum testosterone during the trial. Time to testosterone recovery after last dose of the IMP. Blood samples for analyses of serum testosterone concentrations were collected at Screening and on Days 0 to 126.
Time Frame: Days 56-126
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
days | 46.2 (13.6) | 52.3 (20.6) | 65 (5.7)

5. Secondary Outcome: Profiles of Testesterone Concentration (ng/dL) Following Injections of the Investigational Medicinal Product (IMP)
Description: The PD effects of leuprolide were assessed by measuring serum testosterone concentrations during the trial. The following PD variable was analyzed: The profiles of testosterone concentration (ng/dL) following injections of the IMP. Blood samples for analyses of serum testosterone concentrations were collected at Screening and on Days 0 to 126.
Time Frame: Days 0-126
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
ng/dL
  Day 0 (predose) | 443 [369 to 546] | 321 [269 to 439] | 350 [240 to 465]
  Day 28 (predose) | 20.9 [18.3 to 47] | 24.5 [16.1 to 210] | 18.1 [11.1 to 28.1]
  Day 56 (predose) | 14.6 [10.7 to 19.3] | 13.8 [7.8 to 22] | 12 [9.29 to 15]
  Day 84 | 14.8 [9.17 to 27.6] | 10.6 [7.5 to 18.8] | 12.4 [9.92 to 13.8]
  Day 126 | 423 [258 to 526] | 278 [124 to 470] | 85.8 [16 to 280]

6. Secondary Outcome: Mean Prostate Specific Antigen (PSA) Concentration
Description: The PD effects of leuprolide were assessed by measuring serum PSA concentrations during the trial. The following PD variable was analyzed: PSA (ng/mL) response to IMP. Blood samples for analyses of plasma PSA concentrations were collected at Screening and on Days 0 to 126.
Time Frame: Days 0-126
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Number analyzed (Participants) | 15 | 15 | 17
ng/mL
  Day 0 (predose) | 14.9 [5.8 to 85.4] | 18.8 [9.6 to 93.5] | 14.6 [4.7 to 32.9]
  Day 28 (predose) | 9 [2.8 to 19] | 8.3 [5.9 to 31.5] | 4.6 [2.3 to 8]
  Day 56 (predose) | 3.6 [1.1 to 8.4] | 5.8 [1.1 to 11.2] | 2.1 [0.8 to 4.1]
  Day 84 | 2.3 [1.1 to 5.6] | 2.6 [0.8 to 14] | 1.6 [0.4 to 2.7]
  Day 126 | 4.7 [2.9 to 19.9] | 3.1 [1.5 to 19.1] | 1.6 [0.5 to 3.8]

ADVERSE EVENTS:
Groups:
- CAM2032 3.75 mg: Single subcutaneous buttock injections of CAM2032 3.75 mg on Days 0, 28 and 56.
- CAM2032 7.5 mg: Single subcutaneous buttock injections of CAM2032 7.5 mg on Days 0, 28 and 56.
- Eligard 7.5 mg: Single subcutaneous buttock injections of Eligard 7.5 mg on Days 0, 28 and 56.
Arm/Group | CAM2032 3.75 mg | CAM2032 7.5 mg | Eligard 7.5 mg
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/15 | 0/17
Other Adverse Events (participants affected / at risk) | 14/19 | 12/15 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2032 3.75 mg (N=19) | CAM2032 7.5 mg (N=15) | Eligard 7.5 mg (N=17)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2032 3.75 mg (N=19) | CAM2032 7.5 mg (N=15) | Eligard 7.5 mg (N=17)
Hot flush (Vascular disorders) | 8 (8) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhytmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 3 (6)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (6) | 3 (3) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood urine (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less